CLINICAL TRIAL: NCT01693796
Title: Evaluation of Thyroid Exposure to Radiation Doses During Paediatric Cardiac Catheterisations Performed for Diagnosis or the Treatment of Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A01118-31; 2010-09 (Other: AP HM)
Record Dates: First submitted 2011-04-05; First posted 2012-09-26 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2015-08

CONDITIONS: Cardiac Catheterizations
MeSH Terms: interventions — Blood Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood and urine samples ; Echography

SUMMARY:
The purpose of this study is to determine the average risk for thyroid irradiation for any type of paediatric cardiac catheterization, based on the cummulative at-risk dose of 100 mSv, adjusted to the measured thyroid volume and to the patient's age.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of any patient (< 18 year-old) with congenital heart disease undergoing one or more cardiac catheterization

Exclusion Criteria:

* Exclusion of patients with any type of thyroid dissease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2011-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
exposure to radiation measure | 2 YEARS
  To determine the average risk for thyroid irradiation for any type of paediatric cardiac catheterization, based on the cummulative at-risk dose of 100 mSv, adjusted to the measured thyroid volume and to the patient's age.

SECONDARY OUTCOMES:
exposure to radiation measure | 2 YEARS
  Fit the dose of average irradiation of the thyroid during the catheterizations to the thyroïdien volume

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Chair — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France